CLINICAL TRIAL: NCT06577090
Title: A Phase 2 Study of QW Nimacimab Injection, Compared to Placebo Injection and QW Weekly Nimacimab Injection Co-administered With Semaglutide in Participants Who Are Overweight or Obese
Brief Title: Study to Evaluate the Effect on Obesity of QW Nimacimab and QW Nimacimab Co-administered With Semaglutide vs Placebo
Acronym: CBeyond
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Skye Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBI-018-201
Record Dates: First submitted 2024-08-19; First posted 2024-08-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Nimacimab
MeSH Terms: conditions — Obesity | interventions — semaglutide; Injections

STUDY DESIGN:
Intervention Model Description: Partially blinded combination arm x 2, blinded monotherapy arm x 2, open-label study extension arm monotherapy x 1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants assigned to combination arms will be masked to IP/placebo assignment but unmasked to Wegovy assignment. Participants in the monotherapy arms will remain masked to IP/placebo treatment assignment. Participants who enroll in the study extension (monotherapy arms) will be enrolled into an open-label unblinded 300 mg nimacimab treatment arm. Participants who enroll in the study extension (combination arms) will remain blinded to their treatment assignments with the exception of their Wegovy dose as in the main study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nimacimab injection (Experimental): Nimacimab injection 200 mg
  Interventions: Biological: Nimacimab injection
- Nimacimab placebo injection (Placebo Comparator): Matching nimacimab placebo injection
  Interventions: Biological: Nimacimab placebo injection
- Semaglutide injection + Nimacimab injection 200 mg (Experimental): Semaglutide injection administered according to dose escalation described in semaglutide prescribing information plus concomitant administration of Nimacimab Injection 200 mg
  Interventions: Biological: Nimacimab injection; Combination Product: semaglutide injection
- Semaglutide injection + Nimacimab placebo injection (Active Comparator): Semaglutide injection administered according to dose escalation described in semaglutide Prescribing Information plus concomitant administration of Nimacimab Injection or matching placebo injection
  Interventions: Biological: Nimacimab placebo injection; Combination Product: semaglutide injection
- Open-label 300 mg Nimacimab injection (study extension) (Experimental): Weekly nimacimab injection 300 mg open-label (study extension)
  Interventions: Biological: Nimacimab 300 mg injection

INTERVENTIONS:
Biological: Nimacimab injection — Nimacimab injection 200 mg
  Arms: Nimacimab injection; Semaglutide injection + Nimacimab injection 200 mg
Biological: Nimacimab placebo injection — matching nimacimab placebo injection
  Arms: Nimacimab placebo injection; Semaglutide injection + Nimacimab placebo injection
Combination Product: semaglutide injection — semaglutide injection 0.25 mg, 0.5 mg, 1 mg, 1.7 mg, 2.4 mg + nimacimab 200 mg
  Arms: Semaglutide injection + Nimacimab injection 200 mg; Semaglutide injection + Nimacimab placebo injection
Biological: Nimacimab 300 mg injection — Nimacimab injection 300 mg
  Arms: Open-label 300 mg Nimacimab injection (study extension)

SUMMARY:
This is a proof-of-concept study to assess the safety and efficacy of Nimacimab Injection compared to an active and placebo injection control.

DETAILED DESCRIPTION:
The purpose of this study is to measure the change in body weight with once weekly doses of Nimacimab Injection compared with placebo injection and once weekly Nimacimab Injection co-administered with commercially available semaglutide injection (Wegovy®) in participants with obesity or are overweight with weight-related comorbidities. A study extension has been added to include additional 26 weeks of treatment and 13 weeks of follow up for qualifying participants starting May2025.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Participants must be at least 18 years of age or the legal age of consent in the jurisdiction in which the study is taking place to 65 years, inclusive, at the time of signing the informed consent.
3. Male, female, and/or nonbinary participants.
4. Have Body Mass Index (BMI) of

   1. ≥ 30 kg/m2 to ≤ 45 kg/m2 OR
   2. ≥ 27 kg/m2 and < 30 kg/m2 with clinically confirmed diagnosis of at least 1 of the following weight-related co-morbidities:

   i. dyslipidemia: on lipid-lowering medication or having low-density lipoprotein (LDL) ≥ 160 mg/dL (4.1 mmol/L) or triglycerides ≥ 150 mg/dL (1.7 mmol/L) or high-density lipoprotein (HDL) < 40 mg/dL (1.0 mmol/L) for men or HDL < 50 mg/dL (1.3 mmol/L) for women at screening.

   ii. cardiovascular disease: (for example, ischemic cardiovascular disease, New York Heart Association [NYHA] Functional Classification Class I-II heart failure).

   iii. obstructive sleep apnea syndrome (Salzano 2021).

   iv. controlled arterial hypertension with systolic blood pressure (SBP) < 150 mmHg or diastolic blood pressure (DBP) < 90 mmHg.
5. Have an HbA1c <6.5% at screening.
6. Have had a stable body weight for the 3 months prior to screening (no more than 5% body weight gain and/or loss).
7. If on cardiovascular, anti-hypertensive, must be controlled controlled on a stable dose for 3 months prior to randomization.
8. If on hormone replacement therapy, must be on a stable dose for at least 3 months prior to screening, including use of thyroxine.
9. Females of childbearing potential must agree:

   1. to use an approved method of contraception from screening throughout the study and for at least 90 days after the last dose of study drug.
   2. to not donate ova from screening throughout the study and for at least 90 days after the last dose of study drug.
   3. have a negative pregnancy test at screening and Day 0.
10. Male participants who are (hetero) sexually active must agree that he and his partner will each use an approved method of contraception from screening throughout the study and for at least 90 days after the last dose of study drug.
11. Agreement in male participants to not donate sperm from screening throughout the study and for at least 90 days after the last dose of study drug.

Exclusion Criteria:

1. Have any prior diagnosis of type 1 or type 2 diabetes mellitus (T1DM or T2DM, or rare forms of diabetes mellitus).
2. Have at least 1 laboratory value suggestive of diabetes during screening, including 1 or more of HbA1c ≥ 6.5% (48 mmol/mol), fasting serum glucose ≥ 126 mg/dL (7.0 mmol/L), or random glucose ≥ 200 mg/dL (11.1 mmol/L).
3. Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed > 1 year prior to screening).
4. Have obesity induced by other disorders (for example, Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome) or use of systemic corticosteroids or uncontrolled hypothyroidism. (Hypothyroidism on stable treatment is allowed if thyroid stimulating hormone (TSH) measure within the last 3 months of screening is within normal limits).
5. Have had at any time or plan to have endoscopic and/or device-based therapy for obesity including but not limited to the following:

   1. Mucosal ablation,
   2. Gastric artery embolization,
   3. Intragastric balloon, OR
   4. Duodenal-jejunal endoluminal liner
6. Surgery of any kind within 3 months prior to Day 0 (Baseline) with the exception of minor procedures or determined by the Investigator to be clinically relevant for participation in the study, or any planned surgery during the study.
7. Renal impairment as estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, calculated at screening using the recommended method for estimating eGFR in adults from the National Kidney Foundation Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI 2021) equation (Charles 2024).
8. Acute kidney injury or dialysis within the last 3 months prior to the screening visit
9. Current malignancy with the exception of participants with basal cell carcinoma of this skin, suqamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy.
10. Positive results at screening that indicate an active virological infection at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus.
11. Previous organ or bone marrow transplant.
12. History and/or confirmed seizure disorder; reports febrile and/or idiopathic seizures occurring within the past 2 years.
13. Unstable cardiovascular disease as determined by the Investigator or medical history of myocardial infarction or arterial thromboembolic events within 3 months prior to screening or severe or unstable angina, NYHA Class III or IV disease, or a 12-lead ECG showing QTc interval (Fridericia's formula) >450 msec (males) or >470 msec (females), any tachyarrhythmia, pathologic Q waves, or any other abnormality deemed clinically significant in the opinion of the investigator.
14. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participants' participation for the full duration of the study, or is not in the best interest of the participants to participate in the opinion of the Investigator.
15. Have history of any of the following:

    1. Major Depressive Disorder (MDD)
    2. A lifetime history of suicide attempts
    3. Other severe psychiatric disorder(s) (e.g., schizophrenia, bipolar disorder, etc.)
    4. Use of anti-depressant medication
16. Have a Patient Health Questionnaire-9 (PHQ-9) score ≥ 10 at screening and/or Day 0 (Baseline).
17. At screening or Day 0 (Baseline) have any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) or any suicidal behavior in the lifetime or previous month.
18. History or presence of drug abuse (including medicinal and recreational marijuana use) within the 1 year prior to Day 0 (Baseline) or urine drug assay at screening or Day 0 (Baseline) positive (includes: amphetamines, barbiturates, cocaine metabolites, opiates, benzodiazepines, and cannabinoids).
19. Prior exposure to study drugs

    1. Nimacimab injection
    2. Glucagon-like peptide-1 (GLP-1) agonist.
    3. Allergy to active or inactive component of Nimacimab
    4. Allergy to active or inactive component(s) of GLP-1 agonist
20. Female participants who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the study.
21. Aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 × upper limit of normal (ULN) at screening. One repeat test may be allowed within 7 days of the receiving the result, at the discretion of the Investigator.
22. Absolute neutrophil count ≤ 1.5 × 109/L.
23. Platelets ≤ 120 × 109/L.
24. Hemoglobin (Hgb) < 13.5 g/dL in males and < 12 g/dL in females.
25. Currently or have participated in a study of an investigational product or used an investigational device within 12 weeks and/or 5 times the half-life of the investigational product prior to the (Day 0, Baseline) first dose of study treatment.
26. Current use of any medication that is known to cause weight loss or participation in a structured weight loss program within the last 6 months prior to screening
27. Employees of the Sponsor, contract research organization (CO) involved in the conduct of the study, or investigational site, or immediate family members of the employees.
28. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer of 1.5 ounces [45 mL] of hard liquor) within 6 months of screening.

Study Extension Eligibility Criteria

Participants are eligible to be included in the extension only if all the following criteria apply:

1. Completed Week 26 of the Main study including Week 25 on study treatment. Participants who completed Week 26 of the Main study but discontinued study treatment prior to that visit are not eligible to participate.

   1. Participants in the combination arms (Nimacimab Injection or placebo + Semaglutide) of the Main study must roll over within 4 weeks of Main study Week 26
   2. Participants in the monotherapy arms (Nimacimab Injection or placebo) of the Main study can roll over anytime after they have completed Week 26 on study treatment but before completing the 13-week follow-up period.
2. Does not have any condition that interferes with the ability to complete the Extension in the judgment of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight (main study) | From Baseline to Week 26
  Percent of participants who have a reduction in body weight
Nature, frequency and severity of AEs (study extension) | Baseline through Week 38 of study extension (approximately 10 months of participation)
  Nature, frequency and severity of treatment-emergent adverse events, including serious adverse events and adverse events of special interest

SECONDARY OUTCOMES:
Change in body weight (main study) | From Baseline to Week 26
  Change in body weight in kg
Change in waist circumference (main study) | From Baseline to Week 26
  Change in waist circumference in cm
Change in waist circumference (study extension) | From baseline to Week 26 of study extension (approximately 7 months of participation)
  Change in waist circumference in cm
Change in lean versus fat mass ratio measured by DXA (main study) | From Baseline to Week 26
  Change in lean versus fat mass ratio measured by DEXA (DXA) scan.
Change in lean versus fat mass ratio measured by DXA (study extension) | From baseline to Week 26 of study extension (approximately 7 months of participation)
  Change in lean versus fat mass ratio measured by DEXA (DXA) scan.
Change in BMI (main study) | From Baseline to Week 26
  Change in BMI (weight and height will be combined to report BMI in kg/m^2)
Change in BMI (study extension) | From baseline to Week 26 of study extension (approximately 7 months of participation)
  Change in BMI (weight and height will be combined to report BMI in kg/m^2)
Percent of participants with greater than/equal to 5% body weight reduction as well as greater than/equal to 10% body weight reduction (main study) | From Baseline to Week 26
  Percent of participants with specific body weight reduction (percent based on weight measured in kg)
Percent change in body weight (kg) (study extension) | From baseline to Week 26 of study extension (approximately 7 months of participation)
  Change in body weight (percent based on weight measured in kg)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Skye Bioscience, Inc.
Locations (16):
- United States (16):
  - Pinnacle Research Group, Anniston, Alabama
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - ACCEL Research Sites, Atlanta, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - L-MARC Research Center, Louisville, Kentucky
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Palm Research Center, Las Vegas, Nevada
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - Weill Cornell Medicine, New York, New York
  - Accellacare of Wilmington, Wilmington, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Rainier Clinical Research Center, Renton, Washington